CLINICAL TRIAL: NCT05739149
Title: Microvessel Ultrasound Imaging of the Skin and Subcutaneous Tissues to Evaluate Wound Healing in Patients With Chronic Ulcers
Brief Title: A Study to Evaluate Microvessel Ultrasound Imaging of Wound Healing in Patients With Chronic Ulcers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Michael R. Moynagh, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-012021
Record Dates: First submitted 2023-02-13; First posted 2023-02-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Non-Healing Ulcer of Skin; Non-healing Wound; Lower Extremity Wound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Microvessel Ultrasound Imaging for Chronic Ulcers (Experimental): Subjects with chronic diabetic ulcers and venous ulcers will undergo wound debridement and treatment as standard of care and receive research microvessel ultrasound examination and two skin biopsies
  Interventions: Diagnostic Test: Microvessel Ultrasound Examination; Procedure: Skin Biopsy

INTERVENTIONS:
Diagnostic Test: Microvessel Ultrasound Examination — Ultrasound to evaluate microvessel formation and elastography or stiffness of the tissues around the ulcer and in an area of unaffected skin
Procedure: Skin Biopsy — Dermatology will remove a small piece of skin from the affected ulcer area and control skin

SUMMARY:
The purpose of this research is to explore the use of high-resolution microvessel ultrasound imaging system to look for scarring and to monitor wound healing and to see if treatment affects the amount of tiny vessels and circulation around the wound.

ELIGIBILITY:
Inclusion Criteria:

* Chronic wound in the course of diabetic foot ulcers and/or lower extremity venous ulcers with duration of at least 6 weeks and the wound surface not less than 2 sq. cm and not greater than 15 sq. cm, without evidence of active infection of the wound at the time of qualification to participate in the study
* Meets criteria for stalled chronic wound defined as less than 50% reduction in wound size after 30 days of standard of care management.
* For chronic venous ulcers, ultrasound demonstrates venous reflux >0.5 seconds
* Satisfactory blood glucose control - fasting not more than 110 mg%, HbA1c <6.5%
* Satisfactory blood supply to the wound verified by the measurement of the oxygen level of the foot tissue (TCPO2 > 30mmHg) in patients with neuropathic etiology of diabetic foot syndrome
* In the case of the patients with the wounds of ischemic component, the condition for qualification is a clinical improvement of the limb's blood supply as a result of the revascularization procedure documented by ultrasound.
* Ankle-brachial index (ABI) ≥ 0.8

Exclusion Criteria:

* Acute wound with duration less than 6 weeks
* Evidence of active infection or on antibiotics
* Smoker
* For chronic venous ulcers, ultrasound demonstrates venous reflux <0.5 seconds
* Unsatisfactory blood glucose control - fasting more than 110 mg%, HbA1c <6.5%
* Poor blood supply to the wound verified by the measurement of the oxygen level of the foot tissue (TCPO2 < 30mmHg) in patients with neuropathic etiology of diabetic foot syndrome
* Ankle-brachial index (ABI) < 0.
* Pregnancy
* Known allergy to lidocaine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-12-10 (Estimated); Study Completion 2026-12-10 (Estimated)

PRIMARY OUTCOMES:
Microvessel imaging | 3 months
  Number of subject's microvessel imaging results that correlate to the standard of care clinical assessment of wound healing

CONTACTS AND LOCATIONS:
Overall Officials: Michael Moynagh, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Minnesota, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

DOCUMENTS (1):
  • Informed Consent Form (2024-12-11): https://cdn.clinicaltrials.gov/large-docs/49/NCT05739149/ICF_000.pdf